CLINICAL TRIAL: NCT01352598
Title: Phase IV Trial Evaluating the Use of Stereotactic Body Radiotherapy for the Treatment of Prostate Cancer
Brief Title: Stereotactic Body Radiotherapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Jaymeson Stroud, MD, Radiation Oncologist, Mercy Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-022
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; stereotactic radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Body Radiotherapy (Other): Patients will receive 30 - 40 Gy in 4 - 5 fractions. For high risk patients who also receive external beam radiotherapy, the SBRT will be given as 19 - 21 Gy in 2 - 3 fractions.
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — Patients will receive 30 - 40 Gy in 4 - 5 fractions. For high risk patients who also receive external beam radiotherapy, the SBRT will be given as 19 - 21 Gy in 2 - 3 fractions.

SUMMARY:
This study will evaluate the local control rate as well as acute and late toxicity rates of stereotactic body radiotherapy (SBRT) for the treatment of organ confined prostate cancer.

DETAILED DESCRIPTION:
This is a single site, non-randomized, prospective, phase IV trial of patients with organ-confined prostate cancer. Data collected will include patient demographics, pathology data, tumor stage, SBRT dose fractionation scheme, dose received by adjacent critical normal tissues,tumor recurrence data, and acute and late toxicities. Follow up data will be collected during the patient's standard office visits. The anticipated duration of this study is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >= 18 years
* Zubrod performance status of 0-3
* T1-3 N0 M0 adenocarcinoma of the prostate
* Prostate volume ≤ 100 cc
* Signed study-specific consent form

Exclusion Criteria

* Extension of local tumor to involve adjacent organs other than seminal vesicles (T4)
* Prostate volume > 100 cc
* Nodal involvement
* Metastatic disease
* Prior pelvic radiotherapy except as part of combination therapy for prostate cancer
* History of scleroderma
* Patients with psychiatric or addictive disorder that would preclude obtaining informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-06; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Hospital St. Louis, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiotherapy: Patients will receive 30 - 40 Gy in 4 - 5 fractions. For high risk patients who also receive external beam radiotherapy, the SBRT will be given as 19 - 21 Gy in 2 - 3 fractions.
  stereotactic body radiotherapy: Patients will receive 30 - 40 Gy in 4 - 5 fractions.
  For high risk patients who also receive external beam radiotherapy, the SBRT will be given as 19 - 21 Gy in 2 - 3 fractions.
Period: Overall Study
Arm/Group | Stereotactic Body Radiotherapy
Started | 84
Completed | 72
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 61
Age, Continuous [Mean (Full Range); unit: years] | 68 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 66
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 84

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Control Rate
Description: Serial blood tests for prostate specific antigen (PSA) levels will be obtained at regular intervals (every 3 months).The "Phoenix definition" for biochemical recurrence (nadir + 2 ng/ml) will be used. Biochemical control rate will be expressed based on subjects experiencing tumor control (complete, partial, or stable) vs. subjects experiencing disease progression.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 71
Participants
  Complete, partial, or stable tumor control | 71
  Disease progression | 0

2. Secondary Outcome: Late Toxicity Rate
Description: Toxicity will be recorded as a measure of patients who experienced adverse events within 1 year of study treatment.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 74
Participants
  Patients who experienced no adverse events | 68
  Patients who experienced adverse events | 6

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse event and mortality information collection was limited by 12 study subjects that became unavailable or otherwise did not respond during the course of the 5 year follow-up period. 10 of these 12 study subjects did not make follow-up appointments and were not able to be contacted prior to the end of the first year of follow-up. This caused some discrepancy within the number of patients for whom adverse event data and mortality affects and applies to within the record.
Arm/Group | Stereotactic Body Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 1/74
Other Adverse Events (participants affected / at risk) | 5/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiotherapy (N=74)
GU Bleeding (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiotherapy (N=74)
Change in urinary frequency (Renal and urinary disorders) | 4 (4)
Impotence (Reproductive system and breast disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT01352598/Prot_SAP_ICF_000.pdf